CLINICAL TRIAL: NCT02393703
Title: Interrogation of Exosome-mediated Intercellular Signaling in Patients With Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institutes of Health (NIH) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 15-015
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer; Benign Pancreatic Disease
Keywords: exosomes; 15-015
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, pancreatic fluid, and pancreas tissue

SUMMARY:
The purpose of this study is to isolate and analyze exosomes, which are tiny carriers of important proteins and nucleic acids that serve as messenger systems in the blood and tissue. Blood and tissue from patients with pancreatic cancer will be compared with blood and tissue from patients with noncancerous pancreatic disease. Including patients without cancer will allow the investigators to establish "normal" values, which currently do not exist. The investigators will then look to see whether exosome activity has a connection to disease recurrence and outcomes in patients. The results of this study will be the basis for future studies exploring this area.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years of age undergoing pancreaticoduodenectomy, partial or complete pancreatectomy, and duodenal ampullectomy for presumed ductal adenocarcinoma, intraductal papillary mucinous neoplasm (IPMN) or pancreatic neuroendocrine tumors, without an invasive component; or other benign pancreatic disease will be eligible.
* For third part of the study, recipient of neoadjuvant chemotherapy will be accrued to the neoadjuvant group (25 patients). Patients without neoadjuvant chemotherapy will be accrued to the non-neoadjuvant group (25 patients).

Exclusion Criteria:

* The presence of metastatic disease or disease that precludes resection
* For first and second part of the study, receipt of neoadjuvant chemotherapy or radiation for the index cancer within 6 months of being enrolled in the study
* For third part of the study, receipt of neoadjuvant radiation for the index cancer within 6 months of being enrolled in the study
* INR >2
* Known clotting factor deficiency or hypercoagulable state
* Any patient with the need or anticipated need for full anti-coagulation during hospitalization for the resection.
* Receipt of antiplatelet agents (other than aspirin) in the preceding week prior to resection.
* IPMN or pancreatic neuroendocrine tumors by radiographic imaging with high suspicion for invasive component Additionally, if at the discretion of the operating surgeon, blood collection would lead to undue morbidity, the patient will be excluded and replaced

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSKCC clinic
Sampling Method: Non-Probability Sample
Enrollment: 181 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
successful isolation of exosomes | 1 year
  isolation of at least 100,000 microvesicles is needed for exosomes purification for down stream applications such as proteomics and RNA sequencing.

SECONDARY OUTCOMES:
evaluation of the liver microenvironment | 1 year
  for alterations in cellular infiltrate and ECM using IF and IHC

OTHER OUTCOMES:
evaluation of the omental microenvironment | 1 year
  for alterations in cellular infiltrate and ECM using IF and IHC

CONTACTS AND LOCATIONS:
Overall Officials: William Jarnagin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/